CLINICAL TRIAL: NCT02042456
Title: Automated Breast Ultrasound and Digital Breast Tomosynthesis Screening Compared to Full Field Digital Mammography in Women With Dense Breasts
Status: Terminated | Type: Observational
Why Stopped: Change in study staff at the site, change in Sponsor direction
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 124.03-2013-GES-0003
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; dense breasts; mammography screening; Screening techniques; women
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main Cohort: Subjects enrolled in this group will receive a full field digital mammogram, digital breast tomosynthesis exam and an automated whole breast ultrasound exam as part of their visit.
  Interventions: Device: Digital Breast Tomosynthesis; Device: Automated Whole Breast Ultrasound; Device: Full Field Digital Mammography

INTERVENTIONS:
Device: Digital Breast Tomosynthesis — digital breast tomosynthesis technology
  Other Names: GE SenoClaire DBT with V-Preview
Device: Automated Whole Breast Ultrasound — Automated Whole Breast Ultrasound
  Other Names: Invenia ABUS
Device: Full Field Digital Mammography

SUMMARY:
This study is investigating whether automated whole breast ultrasound can improve detection of cancer in breast cancer screening when used as a supplement to mammography or as a supplement to digital breast tomosynthesis

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed declaration of informed consent or have a legally authorized representative provide signed declaration of informed consent for participation in all study procedures;
* Women aged ≥18 years at the time of enrollment;*
* Women with a previous determination of dense breasts determined by mammogram as heterogeneously dense or extremely dense;
* At moderately increased or high risk (>15% lifetime risk) for breast cancer based on meeting one or more of the ACS criteria 1:

AND Referred for screening mammography

Exclusion Criteria:

* Have been screened using any breast imaging technology in <12 months immediately prior to enrollment;
* Exhibit breast cancer symptoms according to assessment by the subject's health care provider within one year prior to enrollment;
* Diagnosed with breast cancer, with or without metastasis, within one year prior to enrollment;
* Are currently pregnant as determined per standard clinical practice at the investigational site;
* Present with contraindications to any imaging examination required in the study protocol;
* Have breast implants; OR
* Are lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the patients arriving at the clinic for yearly breast cancer screening exams
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Abnormal interpretation rate | One Year
  Abnormal interpretation rates for each modality (FFDM and DBT+V-Preview, with and without ABUS+V-Preview).

SECONDARY OUTCOMES:
Sensitivity | One Year
  Sensitivity will be assessed for each imaging modality: FFDM and DBT+V-Preview, with and without ABUS
Specificity | One Year
  Specificity will be assessed for each imaging modality: FFDM and DBT+V-Preview, with and without ABUS
Cancer Rate | One Year
  Cancer Rate will be assessed for each imaging modality: FFDM and DBT+V-Preview, with and without ABUS
Positive Predictive Value | One Year
  Positive Predictive Value will be assessed for each imaging modality: FFDM and DBT+V-Preview, with and without ABUS
Negative Predictive Value | One Year
  Negative Predictive Value will be assessed for each imaging modality: FFDM and DBT+V-Preview, with and without ABUS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Seattle Cancer Care Alliance, Seattle, Washington, United States